CLINICAL TRIAL: NCT02543970
Title: A Confirmatory Study for Evaluation of the Treatment by the Celluma3 of Periorbital Wrinkles
Status: Completed | Type: Observational
Sponsor: BioPhotas (Industry)
Responsible Party: Sponsor
Other Study IDs: RLE-001
Record Dates: First submitted 2015-09-04; First posted 2015-09-09 (Estimated); Last update posted 2015-09-09 (Estimated); Status verified 2015-09

CONDITIONS: Wrinkled Structure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary objective of this study is to confirm the safe and effective use of the Celluma3 for the reduction in the appearance of periorbital wrinkles.

DETAILED DESCRIPTION:
This clinical study is an open label investigation into the use of the Celluma3 for the effective treatment of periorbital wrinkles.

Test subjects will visit a study center for thirty minute treatments, three times per week, for a period of four weeks, and a twelve week post-treatment follow up after the final treatment. Test subjects will have photos taken at the start, at the end of the four week treatment, and at the final twelve week post-treatment follow up visit.

One of the three Clinical Investigators, will act as the Principal Investigator and all three Clinical Investigators will evaluate the test subjects for inclusion and final results. The Clinical Research Associate (CRA) will monitor the study for conformance to the test protocol.

There will be seven estheticians participating in the study and there will be fifty test subjects recruited.

ELIGIBILITY:
Inclusion Criteria:

1. 30-75 years of age
2. Fitzpatrick Skin Color Type I-IV
3. Clinical evidence of mild to moderate facial wrinkles as specified by the Fitzpatrick Classification of Facial Wrinkling (Perioral and Periorbital) for the degree of wrinkling and elastosis.
4. Willingness and ability to comply with the protocol requirements, including returning for follow up visits and abstaining from excluded behaviors for the duration of the study.
5. Willingness and ability to provide written consent for use of photographic record and adherence to photographic procedures (i.e., removal of makeup and jewelry).
6. Willingness and ability to provide written informed consent prior to any study-related procedure.
7. Absence of any of the exclusionary criteria

Exclusion Criteria:

1. Subject who is pregnant, nursing, or planning to become pregnant during the course of the study.
2. Subjects who have any history of diabetes.
3. Subjects who, in the preceding 12 months prior to the study start, have:

   1. Been exposed to hyaluronic acid, or
   2. any other filler, or
   3. injection for cosmetic purposes related to the face, or
   4. undergone any cosmetic procedure for the face, or
   5. had an active cut, wound or infection of the face, or
   6. had oral isotretinon.
4. Subjects who, in the preceding six months prior to the study start, have:

   1. Had any botulinum toxin ("Botox"), or
   2. had ablative skin resurfacing on the glabellar area.
5. Subjects who, in the preceding three months prior to the study start, have:

   1. Had retinoid, microdermabrasion or prescription level glycolic acid treatments, or
   2. had any compromising procedure in the opinion of any clinical evaluator.
6. Any other diagnosis of any contraindication in the current User Manual.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Test subjects will be between the ages of 30-75, Type I-IV Fitzpatrick Skin Color, and willingness and ability to participate and comply with the test protocol and absence of exclusionary criteria.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2015-02; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Reduction of Periorbital Wrinkles | 16 weeks
  4 weeks of treatment and 12 week follow-up post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jesse Mitchell, MD, FAAD, Principal Investigator